CLINICAL TRIAL: NCT00007241
Title: Osteoarthritic Knee Isometric Exerciser for Home Use
Brief Title: Muscle Strengthening Device for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44AR045153 (NIH); NIAMS-053
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2003-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee; OA; Isometric; Exercise; Strengthening; Joint-related pain
MeSH Terms: conditions — Osteoarthritis; Motor Activity

INTERVENTIONS:
Device: Isometric exercise

SUMMARY:
Studies have shown that isometric strengthening helps people with osteoarthritis of the knee. Isometric strengthening is muscle-strengthening exercise without movement, in which a person applies a force against a resistant object--for example, pushing against a brick wall. This study will test the effectiveness of a portable isometric exercise device for home use that guides a person through an exercise program using various forms of feedback. We will look at whether people exercising with the device achieve better outcomes (results) in pain, stiffness, strength, and functional measures compared to people who do not use the device or people exercising according to printed material from arthritis organizations.

DETAILED DESCRIPTION:
Previous studies have shown that isometric strengthening is beneficial in managing osteoarthritis of the knee. This type of exercise can decrease joint-related pain and stiffness while increasing strength and functional measures. However, individuals rarely adhere to isometric exercise for any lengthy period of time because there has not been a way to measure applied force and performance over time in the home setting. In addition, this type of exercise has often been described as "boring." We believe that being able to monitor one's progress is essential in maintaining adherence to an isometric exercise program. This study will examine the effectiveness of a portable isometric exercise device for home use that guides the user through an exercise protocol by means of various forms of feedback.

We hypothesize that individuals exercising with the device will achieve better outcomes in pain, stiffness, strength, and functional measures than a control group or a group exercising according to printed material from arthritis advocacy groups. We will randomly assign study participants meeting eligibility criteria to the exercise device group, exercise according to printed material group, or control group. We will conduct measures in all groups during a clinic visit at baseline, 2, 4, 6, and 8 weeks. As subjects in the exercise device group strengthen their leg muscles, a physical therapist will likely need to adjust upward the target force for different leg positions during every clinic visit, 2 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Able to give conformed consent.
* Age > 18.
* Pain symptoms provoked by activity in the more symptomatic knee of between (and inclusive of) 3/10 and 8/10 on a verbal analog scale.

Exclusion Criteria:

* Participation in a strengthening program of the knees in the past month.
* Uncontrolled or functionally limiting cardiac disease.
* Uncontrolled hypertension.
* Severe peripheral neuropathy (i.e., insensate to the Simmes 5.07 monofilament).
* Knee flexion contracture greater than 10 degrees.
* Intra-articular steroids in the past 3 months, or hyaluronic acid in the last 9 months.
* Poor health that would impair compliance or assessment.
* Arthroscopy of either knee in the past six months.
* Lateral instability of > 15 degrees, or posterio-anterior instability of greater than 1 cm.
* Knee pain due to pes anserine bursitis.
* Active fibromyalgia.
* Active alcohol or substance abuse.
* Arthritis other than osteoarthritis in the more symptomatic knee.
* Pregnancy.
* History of cancer (other than skin cancer) not in remission.
* Symptomatic spine, hip, ankle, or foot disease other than osteoarthritis that would interfere with assessment of the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92
Dates: Start 2001-09; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Kirk A. Reinbold, PhD, Principal Investigator — Preventive Medical Technologies, Inc.
Locations (6):
- United States (6):
  - Clinical Research Consultants, Inc., Trumbull, Connecticut
  - Radiant Research, Inc., Moorestown, New Jersey
  - Rochester Clinical Research, Inc., Rochester, New York
  - Preventive Medical Technologies, Inc., Philadelphia, Pennsylvania
  - Radiant Research, Inc., Wyomissing, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island

REFERENCES:
- [Background] Goldman RJ, Reinbold KA, Iglarsh ZA, Neustadter LM, Oatis CA, Schumacher HR. Phase I design and evaluation of an isometric muscle reeducation device for knee osteoarthritis rehabilitation. J Rehabil Res Dev. 2003 Mar-Apr;40(2):95-107. doi: 10.1682/jrrd.2003.03.0095. PMID 15077636